CLINICAL TRIAL: NCT01585402
Title: An Open-label, Non-Randomized, Single-Arm Pilot Study to Evaluate the Effectiveness of Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Brief Title: Etidronate for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120110; 12-H-0110
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Results first posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2021-08

CONDITIONS: Arterial Calcification; CD73 Deficiency
Keywords: NT5E; Bisphosphonates; Vascular Calcifications; Joint Capsule Calcifications; Inherited Disease
MeSH Terms: conditions — Vascular Calcification; Genetic Diseases, Inborn | interventions — Etidronic Acid; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Etidronate Treatment for Arterial Calcifications due to Deficiency in CD73 (ACDC) (Experimental): Participants diagnosed with Arterial Calcifications due to Deficiency in CD73 (ACDC) will receive Etidronate. Etidronate will be administered orally at total dose of 20mg/kg daily x 14 days, followed by 10 weeks off study drug (12 weeks = one cycle). Participants may receive up to 12 cycles of etidronate.
  Interventions: Drug: Etidronate; Device: MRI Scan

INTERVENTIONS:
Drug: Etidronate — Didronel (etidronate disodium)- Didronel tablets contain either 200 mg or 400 mg of etidronate disodium, the disodium salt of (1-hydroxyethylidene) diphosphonic acid, for oral administration. This compound, also known as EHDP. regulates bone metabolism. It is a white powder, highly soluble in water. The 400 mg tablets are white capsule-shaped tablets with ED 400 on one side and G on the other side.
  Other Names: Etidronate disodium; Didronel
Device: MRI Scan — Visit on day 0 and visit at 36 month - Exploratory MRI studies may be employed to evaluate the lumen of the artery and degree of collateral vessels, given that the high degree of calcification is precluding that evaluation by CT.

SUMMARY:
Background:

* Arterial Calcifications due to Deficiency in CD73 (ACDC) is a rare genetic disease. People with ACDC develop calcification in the arteries of the lower extremities as well as calcium deposit in the joints of the fingers, wrists, ankles and feet. The lower extremities calcification causes claudication because of severe ischemia requiring at time revascularization procedures. the calcium deposits in the joints causes severe debilitating pain in the hands and feet. Currently, there are no standard treatments for ACDC.
* Etidronate is a bisphosphonate that interferes with bone metabolism. It is approved to treat Paget's disease, a condition in which the bones are soft and weak and may be deformed, painful, or easily broken. It is also used to treat high blood calcium levels. Researchers want to see if it can be used to treat the calcifications of ACDC and improve pain and blood flow in the lower extremities and arthritic pain of the hands and feet.

Objectives:

- To see if etidronate is a safe and effective treatment for ACDC.

Eligibility:

- People between 18 and 80 years of age who have been diagnosed with ACDC.

Design:

* Participants will be screened with a physical exam and medical history. They will also have imaging studies, including CT scan of the lower extremities, x-rays and DEXA bone scans, before starting treatment. Blood and urine samples will be collected. An exercise tolerance test will also be given and ABI (ankle brachial index will be measured.
* Participants will take etidronate by mouth once a day for 14 days every 3 months. They will be assigned an individualized 6- month drug schedule to follow.
* Participants will have regular study visits throughout the treatment period. These visits will involve imaging studies, full dental exams, and blood and urine tests. Participants will also have exercise tolerance tests and ABIs measured.
* Participants may also provide tissue samples for further study.
* Treatment will continue for up to 3 years as long as the side effects are not severe and the condition does not become worse. Participants will have a final follow-up visit after stopping treatment.

DETAILED DESCRIPTION:
We have recently identified a novel genetic disease affecting nine known adults in whom de novo vascular calcifications develop in the lower extremity arteries and juxta-articular joint capsules of the fingers, wrists, ankles and feet. This rare disease results from bi-allelic mutations in the gene ecto-5-prime-nucleotidase (NT5E), encoding the CD73 protein. CD73, an enzyme involved in the extracellular ATP metabolic pathway, converts extracellular AMP to adenosine and inorganic phosphate. The clinical symptoms of this rare disease, termed ACDC (Arterial Calcifications due to Deficiency in CD73), include claudication of the calves, thighs, and buttocks, chronic ischemic pain of the feet at rest with threat of potential limb loss, and debilitating rheumatoid pain in the wrists and hands. Radiological and histological evaluations do not resemble classic atherosclerotic vascular calcification, since the calcification and dysplasia in ACDC occur in the medial portion of the arterial blood vessel wall. Data from patient-specific cell lines indicate increased activity of tissue non-specific alkaline phosphatase (TNAP), a key mediator of pathological ectopic tissue calcification, and thus reveals a potential therapeutic target.

To date, no effective therapy exists for ACDC patients. However, since bisphosphonates are potent competitive inhibitors of TNAP activity and are widely used to modulate bone metabolism, they may beneficially alter vascular calcification. In addition, our preliminary in vitro studies demonstrate the effectiveness of etidronate, a nitrogen-containing bisphosphonate, in lowering TNAP activity in cells isolated from ACDC patients. Etidronate, and bisphosphonates in general, have proven safe and are well tolerated by most patients.

This protocol provides for the administration of etidronate to ACDC patients, for whom no alternative treatment is available. Patients will be examined at the NIH Clinical Center bi-annually for 3 years. The primary objective of this clinical study is to test the effectiveness of etidronate in attenuating the progression of lower extremity arterial calcification and vascular blood flow based on CT calcium score and Ankle Brachial Index (ABI).

ELIGIBILITY:
* INCLUSION CRITERIA

Inclusion and exclusion criteria are to be assessed at Screening and Baseline prior to starting study drug. Each subject must meet the following criteria to be enrolled in this study:

* Subjects must be diagnosed with ACDC based on genetic tests confirming mutation(s) in NT5E and evidence of lower extremity arterial calcifications.
* Either gender and any ethnic background or race
* Age 18-80 years
* Willingness and legal ability to give and sign informed study consent
* Willingness to travel to NIH and local sites for scheduled protocol studies and treatment

EXCLUSION CRITERIA

Subjects who meet any of the following criteria will be excluded from the study:

* Subjects not diagnosed with ACDC
* Subjects <18 or >80 years of age
* Subjects who are unable or unwilling to sign an informed consent
* Severe renal impairment (estimated creatinine clearance/eGFR of < 30ml/min calculated using CKD-EPI equation)
* Longstanding diabetes mellitus (more than 10 years)
* Known abnormality of the esophagus that would interfere with the passage of the drug
* Known sensitivity to etidronate
* Pregnancy
* Any other medical or social condition that, in the opinion of the Principal Investigator, might put the subject at risk of harm during the study or might adversely affect the interpretation of the study data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-08-20 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Brofferio, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] St Hilaire C, Ziegler SG, Markello TC, Brusco A, Groden C, Gill F, Carlson-Donohoe H, Lederman RJ, Chen MY, Yang D, Siegenthaler MP, Arduino C, Mancini C, Freudenthal B, Stanescu HC, Zdebik AA, Chaganti RK, Nussbaum RL, Kleta R, Gahl WA, Boehm M. NT5E mutations and arterial calcifications. N Engl J Med. 2011 Feb 3;364(5):432-42. doi: 10.1056/NEJMoa0912923. PMID 21288095
- [Background] Fleisch H. Bisphosphonates: mechanisms of action. Endocr Rev. 1998 Feb;19(1):80-100. doi: 10.1210/edrv.19.1.0325. No abstract available. PMID 9494781
- [Background] Russell RG. Bisphosphonates: mode of action and pharmacology. Pediatrics. 2007 Mar;119 Suppl 2:S150-62. doi: 10.1542/peds.2006-2023H. PMID 17332236
- [Derived] Ferrante EA, Cudrici CD, Rashidi M, Fu YP, Huffstutler R, Carney K, Chen MY, St Hilaire C, Smith K, Bagheri H, Katz JD, Ferreira CR, Gahl WA, Boehm M, Brofferio A. Pilot study to evaluate the safety and effectiveness of etidronate treatment for arterial calcification due to deficiency of CD73 (ACDC). Vasc Med. 2024 Jun;29(3):245-255. doi: 10.1177/1358863X241235669. Epub 2024 Apr 3. PMID 38568107
- [Derived] Snijders BM, Mathijssen G, Peters MJ, Emmelot-Vonk MH, de Jong PA, Bakker S, Crommelin HA, Ruigrok YM, Brilstra EH, Schepers VP, Spiering W, van Valen E, Koek HL. The effects of etidronate on brain calcifications in Fahr's disease or syndrome: rationale and design of the randomised, placebo-controlled, double-blind CALCIFADE trial. Orphanet J Rare Dis. 2024 Feb 7;19(1):49. doi: 10.1186/s13023-024-03039-7. PMID 38326858
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-H-0110.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the National Institutes of Health Clinical Care Center at Bethesda, Maryland from August 2012 to August 2021.
Period: Overall Study
Arm/Group | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Ankle-brachial Index at Rest at Pre-treatment, On-treatment and Post-treatment of Etidronate in Participants Diagnosed With ACDC
Description: Ankle-brachial Index (ABI) at rest at pre-treatment, on-treatment and post-treatment of etidronate in participants diagnosed with ACDC.
  ABI is the ratio of the blood pressure in the lower and upper extremities obtained by dividing the blood pressure in an artery of the ankle by the blood pressure in an artery of the arm. Interpreting ABI values indicate the amount of arterial disease. Interpretation is as follows: > or equal to 1.3 is noncompressible vessel, > or equal to 1.0 is normal, 0.9 to 0.99 is borderline or equivocal, 0.7 to 0.89 is mild arterial disease, 0.5 to 0.69 is moderate arterial disease, and <0.5 is severe arterial disease.
Time Frame: Up to 2 years (pre-treatment), 3 years (on-treatment) and up to 1 year (post-treatment)
Population: One participant received 11 drug cycles (not 12 cycles) due to discontinuation of the drug by the manufacturer. Participants that underwent lower limb revascularization procedures, measurements obtained after the procedure dates were excluded from analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Number analyzed (Participants) | 7
score on a scale
  Left Side Pre-Treatment at Rest | 0.5741 [0.4801 to 0.6681]
  Left Side On-Treatment at Rest | 0.5411 [0.4479 to 0.6342]
  Left Side Post-Treatment at Rest | 0.5222 [0.4254 to 0.6190]
  Right Side Pre-Treatment at Rest | 0.5266 [0.3746 to 0.6785]
  Right Side On-Treatment at Rest | 0.5322 [0.3827 to 0.6817]
  Right Side Post-Treatment at Rest | 0.5771 [0.4122 to 0.7420]

2. Primary Outcome: Ankle-brachial Index After Exercise at Pre-treatment, On-treatment and Post-treatment of Etidronate in Participants Diagnosed With ACDC
Description: Ankle-brachial Index (ABI) after exercise at pre-treatment, on-treatment and post-treatment of etidronate in participants diagnosed with ACDC.
  ABI is the ratio of the blood pressure in the lower and upper extremities obtained by dividing the blood pressure in an artery of the ankle by the blood pressure in an artery of the arm. Interpreting ABI values indicate the amount of arterial disease. Interpretation is as follows: > or equal to 1.3 is noncompressible vessel, > or equal to 1.0 is normal, 0.9 to 0.99 is borderline or equivocal, 0.7 to 0.89 is mild arterial disease, 0.5 to 0.69 is moderate arterial disease, and <0.5 is severe arterial disease.
Time Frame: Up to 2 years (pre-treatment), 3 years (on-treatment) and up to 1 year (post-treatment)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Number analyzed (Participants) | 7
score on a scale
  Left Side Pre-Treatment after Exercise | 0.5658 [0.4651 to 0.6664]
  Left Side On-Treatment after Exercise | 0.5310 [0.4320 to 0.6300]
  Left Side Post-Treatment after Exercise | 0.5031 [0.3989 to 0.6073]
  Right Side Pre-Treatment after Exercise | 0.6056 [0.3927 to 0.8184]
  Right Side On-Treatment after Exercise | 0.5664 [0.3483 to 0.7844]
  Right Side Post-Treatment after Exercise | 0.4077 [0.1878 to 0.6275]

3. Primary Outcome: Computed Tomography Calcium Score of Lower Extremities at Pre-treatment, On-treatment and Post-treatment of Etidronate in Participants Diagnosed With ACDC
Description: Computed tomography (CT) Calcium Score of lower extremities at pre-treatment, on-treatment and post-treatment of etidronate in participants diagnosed with ACDC.
  According to Cleveland Clinic, a calcium score uses CT to detect calcium deposits in the coronary arteries of the heart. A higher coronary calcium score indicates a higher chance of significant narrowing in the coronary arteries and a higher risk of future heart attack. The Calcium Score range is as follows: zero is no evidence of Coronary Artery Disease (CAD), 1-10 is minimal evidence of CAD, 11-100 is mild evidence of CAD, 101-400 is moderate evidence of CAD and over 400 is extensive evidence of CAD. We applied the same concept to the arteries of the lower extremities. ACDC participants have an overwhelming amount of calcification in the lower extremity vasculature therefore their Calcium Scores are all out of range at baseline and during the study period.
Time Frame: Up to 2 years (pre-treatment), 3 years (on-treatment) and up to 1 year (post-treatment)
Population: One participant received 11 drug cycles (not 12 cycles) due to discontinuation of the drug by the manufacturer. Participants that underwent lower limb revascularization procedures, measurements obtained after the procedure dates were excluded from analysis. ACDC participants have an overwhelming amount of calcification in the lower extremity vasculature therefore their Calcium Scores are all out of range at baseline and during the study period.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Number analyzed (Participants) | 7
score on a scale
  Left Lower Extremity Pre-Treatment | 88817 [20615 to 157019]
  Left Lower Extremity On-Treatment | 91454 [23243 to 159664]
  Left Lower Extremity Post-Treatment | 94358 [26166 to 162551]
  Right Lower Extremity Pre-Treatment | 80289 [12355 to 148222]
  Right Lower Extremity On-Treatment | 81641 [13689 to 149592]
  Right Lower Extremity Post-Treatment | 83950 [16206 to 151694]

4. Secondary Outcome: Changes in Hand Joint Calcification Based on Hand X-ray Before and During Etidronate in Participants Diagnosed With ACDC
Description: Changes in hand joint calcification are based on bilateral hand x-ray before and during Etidronate in participants diagnosed with ACDC as a composite score provided by a radiologist measuring calcium deposit volume (mm^3), calcium deposit density and number of calcifications observed in each finger joint. This is a new scoring system created by our team for the research study, so it has never been used before and healthy volunteer data is not available. However, healthy volunteers would be expected to have no joint calcifications in their hands, in sharp contrast with what we observe in ACDC patients. Density is subjectively defined as 0 equals no calcification, 1 equals barely visible, 2 equals visible with faint margins, 3 equals moderately dense and 4 equals fully dense. The range for the hand X-ray calcification score in this cohort was 288 (minimum) to 863 (maximum).
Time Frame: Up to 2 years (pre-treatment), 3 years (on-treatment)
Population: One participant received 11 drug cycles (not 12 cycles) due to discontinuation of the drug by the manufacturer.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Number analyzed (Participants) | 7
score on a scale
  Left Hand Pre-Treatment | 241.16 [148.45 to 333.87]
  Left Hand On Treatment | 275.15 [173.43 to 376.88]
  Right Hand Pre Treatment | 255.77 [119.40 to 392.13]
  Right Hand On Treatment | 360.20 [209.41 to 510.98]

5. Secondary Outcome: Simple Disease Activity Index Score at Pre-treatment, On-treatment and Post-treatment of Etidronate in Participants Diagnosed With ACDC
Description: Simple Disease Activity Index (SDAI) score at pre-treatment, on-treatment and post-treatment of Etidronate in Participants Diagnosed With ACDC.
  The SDAI is a standard rheumatoid arthritis scores that provide treatment outcome measures on patient joint swelling and pain as well as participants ability to perform daily activity tasks. The SDAI is the sum of five parameters: tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity and level of C-Reactive Protein (mg/dl, normal <1 mg/dl). Total score is defined as: remission as less than 3, low disease activity is between 3 to 11, moderate disease activity is between 11 to 26 and high disease activity is greater than 26. Maximum score possible score is 86 with high disease activity.
Time Frame: Up to 2 years (pre-treatment), 3 years (on-treatment) and up to 1 year (post-treatment)
Population: One participant received 11 drug cycles due to discontinuation of the drug by the manufacturer.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Number analyzed (Participants) | 7
score on a scale
  Pre-Treatment | 18.5919 [14.5739 to 22.6099]
  On-treatment | 8.2987 [5.1215 to 11.4759]
  Post-treatment | 5.0098 [1.1502 to 8.8693]

6. Secondary Outcome: Duke Activity Status Index Score at Pre-treatment, On-treatment and Post-treatment of Etidronate in Participants Diagnosed With ACDC
Description: Duke Activity Status Index (DASI) score at pre-treatment, on-treatment and post-treatment of Etidronate in Participants Diagnosed With ACDC.
  The DASI is an assessment tool used to evaluate the functional capacity of patients with cardiovascular disease (CVD), such as coronary artery disease, myocardial infarction, and heart failure. Positive responses are summed up to get a total score, which ranges from 0 to 58.2. Higher scores would indicate a higher functional capacity.
Time Frame: Up to 2 years (pre-treatment), 3 years (on-treatment) and up to 1 year (post-treatment)
Population: One participant received 11 drug cycles (not 12 cycles) due to discontinuation of the drug by the manufacturer.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Number analyzed (Participants) | 7
score on a scale
  Pre-Treatment | 47.2282 [41.0117 to 53.4447]
  On-treatment | 46.6314 [41.8702 to 51.3926]
  Post-treatment | 50.8242 [44.6566 to 56.9917]

7. Secondary Outcome: Peak Metabolic Equivalents (METS) During Treadmill Test at Pre-treatment, On-treatment and Post- Treatment of Etidronate in Participants Diagnosed With ACDC
Description: Peak Metabolic Equivalents (METS) During Treadmill Test at Pre-treatment, On-treatment and Post- treatment of Etidronate in Participants Diagnosed With ACDC
  A symptom-limited treadmill progressive test (Gardner Protocol) with gradual increase in grade will be performed in accordance with standard practice to evaluation exercise capacity and pain on exertion in subjects with decreased peripheral arterial perfusion. This test will use a constant speed of 2 mph and gradual increase in grade of 2% every 2 minutes beginning at 0% grade.
  METS is a measure of how able a person is to tolerate exercise. No scales exists. METS is calculated by = METs x 3.5 x (your body weight in kilograms) / 200 = calories burned per minute.
Time Frame: Up to 2 years (pre-treatment), 3 years (on-treatment) and up to 1 year (post-treatment)
Population: One participant received 11 drug cycles (not 12 cycles) due to discontinuation of the drug by the manufacturer.
Measure: Mean (95% Confidence Interval); unit: Metabolic Equivalents
Arm/Group | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
Number analyzed (Participants) | 7
Metabolic Equivalents
  Left Lower Extremity Pre-Treatment | 6.2514 [5.4057 to 7.0971]
  Left Lower Extremity On-Treatment | 6.2577 [5.4467 to 7.0687]
  Left Lower Extremity Post-Treatment | 6.2888 [5.4060 to 7.1717]
  Right Lower Extremity Pre-Treatment | 6.2514 [5.4057 to 7.0971]
  Right Lower Extremity On-Treatment | 6.2577 [5.4467 to 7.0687]
  Right Lower Extremity Post-Treatment | 6.2888 [5.4060 to 7.1717]

ADVERSE EVENTS:
Time Frame: 37 months
Description: Adverse events will be captured from the start of the first etidronate administration (day 0) until 30 days following the last dose of treatment. Following this period, any observed or volunteered adverse events will NOT be reported or recorded unless they are greater than Grade 1 and deemed possibly, probably or definitely related to a procedure, test or screening examination that was administered as part of this protocol.
Arm/Group | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC)
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC) (N=7)
Stroke (Nervous system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
External iliac artery stenosis (Vascular disorders) | 1 (1)
Jump graft on the bypass area declining function of previous graft (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etidronate Treatment for Arterial Calcifications Due to Deficiency in CD73 (ACDC) (N=7)
Abdominal pain (Gastrointestinal disorders) | 2 (9)
Bloating (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 7 (34)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (21)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (9)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Cholesterol high (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 4 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Premature atrial contractions (Cardiac disorders) | 1 (1)
Left atrial enlargement; Incomplete right bundle branch block (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 3 (4)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Vivid dreams (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Allergic reaction (Immune system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 2 (3)
Weight loss (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Calcaneus spur (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint inflammation/pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Cold symptoms (Infections and infestations) | 1 (1)
Streptococcus pyogenes (Infections and infestations) | 1 (1)
Strep agalactiae Urinary tract infection (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (2)
Malaise (General disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (5)
Dysgeusia (Nervous system disorders) | 3 (7)
Headache (Nervous system disorders) | 3 (9)
Memory impairment (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 1 (2)
Elevated urine phosphorus (Renal and urinary disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (9)
Left inguinal hernia surgery (General disorders) | 1 (1)
Arthralgia flare swelling of right hand (General disorders) | 1 (1)
Arthralgia flare swelling of right wrist (General disorders) | 1 (1)
Swelling of finger on fourth MCP of right hand (General disorders) | 1 (1)
Hemorrhoids (General disorders) | 1 (2)
Injection site reaction (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Blister on right 4th toe (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (3)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Flu like symptoms (General disorders) | 3 (5)
Hypertension (Vascular disorders) | 2 (5)
Hypotension (Vascular disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT01585402/Prot_SAP_000.pdf